CLINICAL TRIAL: NCT03684031
Title: Impact of Cognitive Control Training on Anger Symptoms and Reactive Aggression (Anger Study)
Brief Title: Impact of Cognitive Control Training on Anger Symptoms and Reactive Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Monique Tremblay, Monique D Tremblay, M.A Ryerson University, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anger Study 2
Record Dates: First submitted 2018-09-22; First posted 2018-09-25 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Anger
Keywords: Reactive Aggression; Anger; Cognitive Control Training; Anger Rumination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Control Training (Experimental): Participants in this arm will complete a computer-based training program two times in the lab. Participants will complete the first training session in the lab during their initial visit and they will return to the lab one week later to complete the second session.
  Interventions: Behavioral: Cognitive Control Training
- Sham Cognitive Control Training Program (Sham Comparator): Participants in this arm will complete a sham training program two times in the lab. The program will look similar in length and design to the experimental training program, but the content of the program will remain affectively neutral. As in the experimental condition, participants will complete the first training session in the lab during their initial visit and they will return to the lab one week later to complete the second session.
  Interventions: Behavioral: Sham Cognitive Control Training Program

INTERVENTIONS:
Behavioral: Cognitive Control Training — A computer-based flanker task that aims to reinforce the recruitment of cognitive control in the presence of hostile/aggressive stimuli.
  Arms: Cognitive Control Training
Behavioral: Sham Cognitive Control Training Program — A placebo version of the computer-based cognitive control training. Designed to appear similar to the experimental task, but will not reinforce the recruitment of cognitive control in the presence of hostile/aggressive stimuli.
  Arms: Sham Cognitive Control Training Program

SUMMARY:
High trait anger is a personality construct characterized by elevations in the frequency, duration, and intensity of anger episodes. According to many social cognitive theories, hostile interpretations of everyday situations contribute to the development and maintenance of anger symptoms. This study will examine the effectiveness of a computer-based cognitive control training task.

DETAILED DESCRIPTION:
Difficulties with anger control are reported in a number of psychological conditions and are associated with social problems, such as dating violence and workplace violence. High trait anger is a personality construct characterized by elevations in the frequency, duration, and intensity of anger episodes. However, the cognitive processes contributing to high trait anger are still poorly understood. According to the Integrative Cognitive Model of Anger and Reactive Aggression (ICM), three cognitive processes jointly contribute to the experience of high trait anger and reactive aggression: 1) hostile interpretation biases; 2) cognitive control; and 3) anger rumination. The proposed study will evaluate the validity of this model in relation to cognitive control using a computer-based cognitive control training (CCT) program.

ELIGIBILITY:
Inclusion Criteria:

1. Score of 22 or higher on the Trait Anger Scale.

Exclusion Criteria:

1. Reports currently receiving psychological treatment or counseling for anger management difficulties.
2. Reports changes in psychiatric medication within the last month.
3. Endorsement of current psychosis or bipolar disorder symptoms.
4. Indicates poor English language proficiency.
5. Reports clinically significant suicidal ideation, intent, or plan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
State-Trait Anger Expression Inventory 2nd Edition | Administered two times over the course of one week. Changes will be examined from visit 1 (before CCT training program) to visit 2 (after CCT training program)
  A self-report measure of the experience of anger.
Computer-based cognitive control assessment | Administered two times over the course of one week. Changes will be examined from visit 1 (before CCT training program) to visit 2 (after CCT training program)
  A behavioural measure of hostility-primed cognitive control involving aggressive and neutral words.

SECONDARY OUTCOMES:
Anger Rumination Scale | Administered two times over the course of one week. Changes will be examined from visit 1 (before CCT training program) to visit 2 (after CCT training program)
  A self-report measure of the degree to individuals focus on experiences with anger. The scale is comprised of four subscales, angry after thoughts (e.g., "Whenever I experience anger, I keep thinking about it for a while"), angry memories (e.g., "I re-enact the anger episode in my mind after it has happened"), understanding causes (e.g., "When someone provokes me, I keep wondering why this should have happened to me"), and thoughts of revenge (e.g. "I have difficulty forgiving people who have hurt me."). Participants will be asked to read each item and rate it in terms of how well it reflects their experience on a 4-point scale from 1 ("almost never") to 4 ("almost always"). Totals for each sub scale will be summed to produce a total score (range: 19-76), with higher scores indicating a greater propensity for rumination.
Depression and Anxiety Stress Scale-21 (DASS-21) | Administered two times over the course of one week. Changes will be examined from visit 1 (before CCT training program) to visit 2 (after CCT training program)
  A self-report measure of depression, anxiety, and stress symptoms.Items are summed for each subscale to create subscale totals (i.e., depression, anxiety, and stress), with higher scores reflecting more severe emotional distress. Symptom score ranges include: normal (0-4), mild (5-6), moderate (7-10), severe (11-13), and extremely severe (14+).
Dot probe task | Administered two times over the course of one week. Changes will be examined from visit 1 (before CCT training program) to visit 2 (after CCT training program)
  A behavioural measure of attentional bias towards angry faces.
Adult Temperament Questionnaire (Effortful Control section) | Administered two times over the course of one week. Changes will be examined from visit 1 (before CCT training program) to visit 2 (after CCT training program)
  A self-report measure of one's ability to suppress inappropriate approach behavior, to perform an action when there is a strong tendency to avoid it, and to shift or focus behaviour.
Reactive-Proactive Aggression Questionnaire | Administered two times over the course of one week. Changes will be examined from visit 1 (before CCT training program) to visit 2 (after CCT training program)
  A self-report measure of an individual's propensity for reactive aggression.
Taylor Aggression Paradigm | Administered one time over the course of one week. Participants will be exposed to the paradigm following the second training session.]
  A behavioural measure of reactive aggression.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The results of this study will be disseminated through conference presentations, journal publications, and through the lab website. Anonymized aggregate participant data may be made available upon request to a publishing journal or individual research group. However, research groups interested in accessing anonymized data will be required to submit a proposal detailing their intended use of the data. Their qualifications will be reviewed based on their proposal and CVs. Individual research groups approved for access will be required to agree to not attempt to re-identify participants, not further distribute data, and not use the data for purposes other than specified in their original proposal. No individual data will be shared.

REFERENCES:
- [Background] Wilkowski BM, Robinson MD. The cognitive basis of trait anger and reactive aggression: an integrative analysis. Pers Soc Psychol Rev. 2008 Feb;12(1):3-21. doi: 10.1177/1088868307309874. Epub 2007 Dec 18. PMID 18453470